CLINICAL TRIAL: NCT04918771
Title: Multicenter Double Blind Placebo-controlled Parallel-group Randomized Clinical Study of Efficacy and Safety of Raphamin in the Treatment of Acute Respiratory Viral Infection in Children Aged 12-18 Years Old
Brief Title: Clinical Study of Efficacy and Safety of Raphamin in the Treatment of ARVI in Children 12-18 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-407-003
Record Dates: First submitted 2021-05-21; First posted 2021-06-09 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-08

CONDITIONS: Acute Respiratory Viral Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raphamin (Experimental): Tablet for oral use.
  Interventions: Drug: Raphamin
- Placebo (Placebo Comparator): Tablet for oral use.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raphamin — Oral administration - not with food. Keep the tablet in the mouth until it is completely dissolved.
  On the 1st day of treatment, 8 tablets are taken according to the following scheme: 1 tablet every 30 minutes in the first 2 hours (a total of 5 tablets in 2 hours), then during the same day, take another 1 tablet 3 times at regular intervals. On the 2nd day and then take 1 tablet 3 times a day. The duration of treatment is 5 days.
  Arms: Raphamin
Drug: Placebo — Oral administration - not with food. Placebo using Raphamin scheme.
  Arms: Placebo

SUMMARY:
The multicenter double-blind placebo-controlled randomized in parallel-group. The objective of this study is to evaluate efficacy and safety of Raphamin in the treatment of acute respiratory viral infection (ARVI) in children aged 12-18 years old.

DETAILED DESCRIPTION:
Design: a multicenter, double-blind, placebo-controlled, parallel-group randomized clinical trial.

The study will enroll outpatient subjects of either gender aged 12-18 old years with clinical manifestations of acute respiratory viral infection (ARVI) within the first days after the onset of the disease. The patients will be recruited during seasonal ARVI morbidity. Collection of history, thermometry, objective examination, laboratory tests, recording concomitant therapy will be made after parent/adoptive parent signing information sheet and informed consent form for the child participation in the clinical study, for children ≥14 years old after signing patient information sheet and informed consent form for children ≥14 years old to participate in the clinical study. The severity of ARVI symptoms will be evaluated with a 4-point scale.

The nasopharyngeal swabs for PCR diagnosis and verification of respiratory viruses will be performed prior to therapy to confirm the viral etiology of ARVI. To rule out the infection caused by the new coronavirus COVID-19 (Coronavirus disease 2019), a rapid test for SARS-CoV-2 antigen will be made. In case of a positive SARS-CoV-2 test, the physician will act in accordance with the current version of the RF MoH Temporary methodological recommendations "Prevention, diagnosis, and therapy of new coronavirus infection (COVID-19)".

If a patient meets all inclusion criteria and does not have any exclusion criteria, at Visit 1 (Day 1), he/she will be randomized into one of two groups: patients of group 1 will take Raphamin according to the dosage regimen for 5 days; patients of group 2 will take Placebo using Raphamin 5-day regimen.

The study will use an electronic patient diary (EPD) for recording morning and evening axillary body temperature (using a classic mercury-free thermometer) and disease symptoms (Symptom Severity Score). Besides, antipyretic dosing (if applicable) and any deterioration in a patient's condition (if applicable, for safety evaluation/AE documentation) will also be recorded in a patient diary. The investigator will provide instructions on filling the diary. At Visit 1 the parent/adoptive parent together with an investigator will record ARVI symptom severity and body temperature in the diary.

Patients will be observed for 14 days (screening, randomization - up to 1 day, treatment period - 5 days, follow-up - up to 2 days; deferred "phone visit" - day 14).

During the treatment and follow-up period the patients/physicians will make 3 visits and the fourth "phone visit" will be scheduled additionally: 1) visits by physician/patient - on Days 1, 5, and 7 (Visits 1, 2, and 3) - in a study center or at home; 2) "phone visit" (Visit 4) - on Day 14.

At Visits 2 and 3, the investigator will perform an objective examination, document changes in the symptoms and concomitant medications, and check patient diaries. At Visit 3 laboratory tests will be performed and compliance will be checked.

"Phone visit" will be performed to interview parents/adoptive parents about the patient's condition, presence/absence of secondary bacterial/viral complications, and use of antibiotics.

During the study, symptomatic therapy and therapy for their co-morbidities are allowed with the exception of the drugs indicated in the section "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender aged 12 to 18 years.
2. Diagnosis of ARVI based on medical examination: axillary temperature ≥ 37.8°C at examination + non-specific flu-like symptoms score ≥4, nasal/throat/chest symptom score ≥2.
3. The first 24 hours after ARVI onset.
4. Contraceptive measures by sexually active adolescents of both genders during the study.
5. Patient information sheet (informed consent form) signed by one parent/adoptive parent of the patient and there is also a signed patient information sheet (informed consent form) for children aged 14 and over.

Exclusion Criteria:

1. Clinical symptoms of severe influenza/ARVI requiring hospitalization.
2. Positive SARS-CoV-2 (COVID-19/Coronavirusdisease2019) antigen test.
3. Suspected pneumonia, bacterial infection (including otitis media, sinusitis, urinary tract infection, meningitis, sepsis, etc.) requiring administration of antibiotics from the first day of illness.
4. Suspected initial manifestations of diseases with symptoms similar to ARVI at onset (other infectious diseases, flu-like syndrome at the onset of systemic connective tissue diseases, and other pathology).
5. Patients requiring antiviral medication prohibited within the study.
6. Medical history of primary and secondary immunodeficiency.
7. Medical history/suspicion of oncology of any localization (except for benign neoplasms).
8. Aggravation or decompensation of chronic diseases (diabetes mellitus, infantile cerebral paralysis, cystic fibrosis, primary ciliary dyskinesia, bronchopulmonary dysplasia, respiratory and ENT congenital defects, etc.) affecting a patient's ability to participate in the clinical trial.
9. Malabsorption syndrome, including congenital or acquired lactase or other disaccharidase deficiency, galactosemia.
10. Allergy/ hypersensitivity to any component of the study drugs used in the treatment.
11. Pregnancy. Breast-feeding.
12. Use of medications specified in the section "Prohibited Concomitant Therapy" within two weeks prior to inclusion in the study.
13. Patients whose parents/adopters, from the investigator's point of view, will not comply with the observation requirements during the study or follow the procedure for taking the study drugs.
14. Medical history of mental diseases of the patient or their parent(s)/adoptive parents.
15. Participation in other clinical trials for 3 months prior to enrollment in this study.
16. Patient's parents/adopters who are related to any of the on-site research personnel directly involved in the study or are an immediate relative of the investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
17. The patient's parent/adopter who work for OOO "NPF "MATERIA MEDICA HOLDING" (i.e. the company's employees, temporary contract workers, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 435 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- Russia (29):
  - Kazan State Medical University, Kazan'
  - Llc "Medlight", Kazan'
  - Specialized Clinical Hospital for Infectious Diseases, Krasnodar
  - Llc "Olla-Med", Moscow
  - Russian National Research Medical University named after N.I. Pirogov, Moscow
  - Morozovskaya Children's City Clinical Hospital of the Moscow Department of Health, Moscow
  - Federal Scientific and Clinical Center for Physical and Chemical Medicine of the Federal Medical and Biological Agency, Moscow
  - Llc "Diagnostics and Vaccines", Moscow
  - Novosibirsk State Medical University, Novosibirsk
  - City Children's Clinical Polyclinic # 5, Perm
  - LLC "Professorial Clinic", Perm
  - Clinical and diagnostic center "Health" of the city of Rostov-on-Don, Rostov-on-Don
  - Children's City Hospital #1 of Rostov-on-Don city, Rostov-on-Don
  - Rostov State Medical University, Rostov-on-Don
  - Ryazan State Medical University named after academician I.P. Pavlov, Ryazan
  - Children's city polyclinic # 44, Saint Petersburg
  - LLC "Energy of health", Saint Petersburg
  - Children's city polyclinic # 35, Saint Petersburg
  - Research Institute of Influenza named after A.A. Smorodintsev, Saint Petersburg
  - Samara Regional Children's Clinical Hospital named after N.N. Ivanova, Samara
  - National Research Mordovian State University named after N.P. Ogarev, Saransk
  - LLC "DNA Research Center", Saratov
  - Smolensk State Medical University, Smolensk
  - Bashkir State Medical University/Department of Outpatient and Emergency Pediatrics, Ufa
  - Volgograd State Medical University/Department of Pediatrics and Neonatology, Volgograd
  - Yaroslavl State Medical University/Department of Pediatrics IPGE, Yaroslavl
  - Yaroslavl State Medical University/Department of Pediatrics № 2, Yaroslavl
  - Clinical Hospital # 2, Yaroslavl
  - LLC "European Medical Center "UMMC-Health", Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 435 patients signed informed consent, of which 10 patients did not pass screening (not meet inclusion criteria or non-inclusion criteria). 5 patients had significant deviations from the procedure for signing informed consent. However, they were randomized and received study therapy. But these patients are not counted as randomized.
Groups:
- Raphamin: Tablet for oral use.
  Raphamin: Oral administration - not with food. Keep the tablet in the mouth until it is completely dissolved.
  On the 1st day of treatment, 8 tablets are taken according to the following scheme: 1 tablet every 30 minutes in the first 2 hours (a total of 5 tablets in 2 hours), then during the same day, take another 1 tablet 3 times at regular intervals. On the 2nd day and then take 1 tablet 3 times a day. The duration of treatment is 5 days.
Period: Overall Study
Arm/Group | Raphamin | Placebo
Started | 206 | 214
Completed | 199 | 205
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Incorrect inclusion ineligible patient | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raphamin | Placebo | Total
Number analyzed (Participants) | 199 | 205 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.7) | 14.2 (1.7) | 14.2 (1.7)
Age, Customized [Count of Participants; unit: Participants]
  12 to 18 years | 199 | 205 | 404
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 107 | 207
  Male | 99 | 98 | 197
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 199 | 205 | 404

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Acute Respiratory Viral Infection (ARVI) Symptoms (ARVI, Confirmed by Polymerase Chain Reaction (PCR)).
Description: Outcome Measure is evaluated on the basis of ARVI, confirmed by Polymerase chain reaction (PCR), i.e virus detection.
  ARVI's resolution criteria: temperature ≤37.3°С + total symptom score (TSS) ≤2. Axillar temperature, 6 flu-like nonspecific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness) and 7 nasal/throat/chest symptoms (runny nose, nasal congestion, sneezing, hoarseness, sore throat, cough, pain/heaviness in chest) were registered for TSS according to the 4-point scale for each of them (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). To calculate TSS absolute axillar temperature (in degrees Celsius) was converted to relative units (or points) using the following scale: ≤37.3 С=0 points; 37.4-38.0 С=1 point; 38.1-39.0 С=2 points; ≥39.1 С=3 points. So the range of TSS was from "0" to "42". The TSS higher score is the worse outcome.
Time Frame: 14 days of observation
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 122 | 107
day | 3.3 (1.7) | 4.4 (2.6)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Mean time to resolution of ARVI symptoms; Test type: Superiority; p = 0.0003, t-test, 2 sided; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [0.51 to 1.67]

2. Secondary Outcome: Severity of ARVI (Clinically Diagnosed and/or PCR-confirmed).
Description: The outcome measure is based on the area under the curve (AUC) for the TSS (Total symptoms score).
  TSS is calculated as a sum of scores for 14 different symptoms. 13 of them are different ARVI manifestations, each of them is evaluated on a scale: 0 (none), 1 (mild), 2 (moderate), 3 (severe). 14th symptom is body temperature (temp) which is converted to its score using following rules:
  if temp <= 37.3 then score = 0 (none) if 37.3 < temp <= 38.0 then score = 1 (mild) if 38.0 < temp <= 39.0 then score = 2 (moderate) if 39.0 < temp then score = 3 (severe) So it is 14 symptoms and the score for each of them varies between 0 and 3. Minimum TSS is 0, maximum is 42 (higher TSS score is worse). AUC is calculated for all timepoints available for patient.
Time Frame: Day1 through Day6 of the treatment and observation
Population: Two subpopulations were analysed:
  1. Patients with clinically diagnosed and/or PCR-confirmed ARVI.
  2. Patients with PCR-confirmed ARVI strictly.
Measure: Mean (Standard Deviation); unit: scores on a scale*days
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 199 | 205
scores on a scale*days
  Severity of ARVI (Clinically Diagnosed and/or PCR-confirmed), AUC score | 44.6 (23.8) | 46.9 (24.3)
  Severity of ARVI (PCR-confirmed), AUC score: number analyzed (Participants) | 122 | 107
  Severity of ARVI (PCR-confirmed), AUC score | 48.3 (25.2) | 53.6 (25.6)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Mean AUC score for severity of ARVI (Clinically Diagnosed and/or PCR-confirmed); Test type: Superiority; p = 0.3274, t-test, 2 sided; Mean Difference (Final Values) = 2.35, 95% CI 2-sided [-2.36 to 7.06]
Statistical Analysis 2: Comparison: Raphamin vs Placebo; Mean AUC score for severity of ARVI (PCR-confirmed); Test type: Superiority; p = 0.1171, t-test, 2 sided; Mean Difference (Final Values) = 5.30, 95% CI 2-sided [-1.34 to 11.93]

3. Secondary Outcome: Percentage of Patients With Resolution of ARVI Symptoms (Clinically Diagnosed and/or PCR-confirmed).
Description: ARVI's resolution criteria: temperature ≤37.3°С + total symptom score (TSS) ≤2. Axillar temperature, 6 flu-like nonspecific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness) and 7 nasal/throat/chest symptoms (runny nose, nasal congestion, sneezing, hoarseness, sore throat, cough, pain/heaviness in chest) were registered for TSS according to the 4-point scale for each of them (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). To calculate TSS absolute axillar temperature (in degrees Celsius) was converted to relative units (or points) using the following scale: ≤37.3 С=0 points; 37.4-38.0 С=1 point; 38.1-39.0 С=2 points; ≥39.1 С=3 points. So the range of TSS was from "0" to "42". The TSS higher score is the worse outcome.
Time Frame: 14 days of observation
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 199 | 205
Participants
  Day 2 | 24 | 16
  Day 3 | 64 | 46
  Day 4 | 96 | 94
  Day 5 | 149 | 136
  Day 6 | 174 | 162
  Day 7 | 191 | 181
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Time to Resolution of ARVI Symptoms (Clinically Diagnosed and/or PCR-confirmed).
Description: as for outcome 3
Time Frame: 14 days of observation
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 199 | 205
day | 3.4 (1.8) | 3.9 (2.4)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; The mean time to Resolution of ARVI Symptoms was analysed; Test type: Superiority; p = 0.0073, t-test, 2 sided; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [0.16 to 1.00]

5. Secondary Outcome: Percentage of Patients With Resolution of ARVI Symptoms (PCR-confirmed).
Description: Outcome Measure is based on the Percentage of Patients With Resolution of ARVI, confirmed by Polymerase chain reaction (PCR), i.e virus detection.
  ARVI's resolution criteria: temperature ≤37.3°С + total symptom score (TSS) ≤2. Axillar temperature, 6 flu-like nonspecific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness) and 7 nasal/throat/chest symptoms (runny nose, nasal congestion, sneezing, hoarseness, sore throat, cough, pain/heaviness in chest) were registered for TSS according to the 4-point scale for each of them (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). To calculate TSS absolute axillar temperature (in degrees Celsius) was converted to relative units (or points) using the following scale: ≤37.3 С=0 points; 37.4-38.0 С=1 point; 38.1-39.0 С=2 points; ≥39.1 С=3 points. So the range of TSS was from "0" to "42". The TSS higher score is the worse outcome.
Time Frame: 14 days of observation
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 122 | 107
Participants
  Day 2 | 16 | 4
  Day 3 | 36 | 16
  Day 4 | 59 | 39
  Day 5 | 95 | 64
  Day 6 | 107 | 77
  Day 7 | 119 | 89
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Dosing Frequency of Antipyretics.
Description: Outcome Measure is based on the rates of antipyretic use per patient during days 1 to 3 of therapy according to the electronic patient diary.
Time Frame: 3 days of therapy
Measure: Mean (Standard Deviation); unit: number of doses
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 199 | 205
number of doses
  Day 1 | 0.43 (0.72) | 0.39 (0.72)
  Day 2 | 0.22 (0.61) | 0.25 (0.66)
  Day 3 | 0.09 (0.38) | 0.07 (0.31)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Dosing Frequency of Antipyretics. Comparison for Day 1; Test type: Superiority; p = 0.3627, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Raphamin vs Placebo; Dosing Frequency of Antipyretics. Comparison for Day 2; Test type: Superiority; p = 0.5578, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Raphamin vs Placebo; Dosing Frequency of Antipyretics. Comparison for Day 3; Test type: Superiority; p = 0.7688, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percentage of Patients Reporting Worsening of Illness.
Description: Outcome Measure is based on the rates of Complications that require the use of antibiotics or hospitalization.
Time Frame: Day 4 through day 14 of the treatment and observation period
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 199 | 205
Participants | 1 | 0
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.4926, Fisher Exact

8. Secondary Outcome: Occurrence and Type of Adverse Events (AE) During the Treatment. AE Severity.
Description: 1. The intensity (severity) of adverse events.
  2. Causal relationship of AEs to the sudy drug.
  3. Outcome of AEs. Based on medical records.
Time Frame: 14 days of observation
Measure: Number; unit: number of cases
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 206 | 214
number of cases
  Severity/Mild | 2 | 6
  Severity/Moderate | 5 | 0
  Causal relationship/Not connected | 7 | 6
  Outcome/Recovery | 6 | 5
  Outcome/Unknown | 1 | 1
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Comparison of severity distributions; Test type: Superiority; p = 0.021, Fisher Exact
Statistical Analysis 2: Comparison: Raphamin vs Placebo; Comparison for outcome distribution; Test type: Superiority; p = 1.00, Fisher Exact

9. Secondary Outcome: Changes in Vital Signs: Pulse Rate/Heart Rate in Beats Per Minute (Bpm).
Description: The outcome measure is based on the medical records. The patient's heart rate (heart rate) is measured by the physician in every visit (on days 1, 5, and 7).
Time Frame: Day 1 through day 7 of the treatment and observation period.
Population: Only non-missing values were analyzed, so numbers analyzed are a bit lower then overall number of participants for visits 2 and 3.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 206 | 214
beats per minute
  Visit 1 | 87.1 (11.4) | 87.2 (10.6)
  Visit 2: number analyzed (Participants) | 201 | 210
  Visit 2 | 77.9 (7.1) | 78.1 (7.2)
  Visit 3: number analyzed (Participants) | 200 | 210
  Visit 3 | 76.3 (7.0) | 76.7 (6.8)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Comparison for Visit 1; Test type: Superiority; p = 0.7848, Median test
Statistical Analysis 2: Comparison: Raphamin vs Placebo; Comparison for Visit 2; Test type: Superiority; p = 0.9596, Median test
Statistical Analysis 3: Comparison: Raphamin vs Placebo; Comparison for Visit 3; Test type: Superiority; p = 0.6902, Median test

10. Secondary Outcome: Changes in Vital Signs: Respiration Rate/Breathing Rate in Breaths Per Minute.
Description: Outcome Measure is based on the medical records. The patient's respiration rate (breathing rate) is measured by physician in every visit (on days 1, 5, and 7).
Time Frame: Day 1 through day 7 of the treatment and observation period.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 206 | 214
breaths per minute
  Visit 1 | 20.8 (3.3) | 20.7 (2.8)
  Visit 2: number analyzed (Participants) | 201 | 210
  Visit 2 | 18.4 (1.9) | 18.6 (1.7)
  Visit 3: number analyzed (Participants) | 200 | 210
  Visit 3 | 18.0 (1.7) | 18.2 (1.7)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Comparison for Visit 1; Test type: Superiority; p = 0.3266, Median test
Statistical Analysis 2: Comparison: Raphamin vs Placebo; Comparison for Visit 2; Test type: Superiority; p = 0.0930, Median test
Statistical Analysis 3: Comparison: Raphamin vs Placebo; Comparison for Visit 3; Test type: Superiority; p = 0.2308, Median test

11. Secondary Outcome: Changes in Vital Signs: Blood Pressure in Units of Millimeters of Mercury (mmHg).
Description: Outcome Measure is based on the medical records. The patient's blood pressure is measured by the physician in every visit (on days 1, 5, and 7).
Time Frame: Day 1 through day 7 of the treatment and observation period.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 206 | 214
mmHg
  Visit 1/Systolic blood pressure | 112 (9.9) | 112 (8.9)
  Visit 2/Systolic blood pressure: number analyzed (Participants) | 201 | 210
  Visit 2/Systolic blood pressure | 111 (9.8) | 112 (8.7)
  Visit 3/Systolic blood pressure: number analyzed (Participants) | 200 | 210
  Visit 3/Systolic blood pressure | 111 (10.2) | 111 (9.4)
  Visit 1/Diastolic blood pressure | 70.0 (5.7) | 69.8 (5.8)
  Visit 2/Diastolic blood pressure: number analyzed (Participants) | 201 | 210
  Visit 2/Diastolic blood pressure | 69.7 (5.7) | 69.5 (5.4)
  Visit 3/Diastolic blood pressure: number analyzed (Participants) | 200 | 210
  Visit 3/Diastolic blood pressure | 69.6 (5.7) | 69.4 (5.9)
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Comparison for Visit 1/Systolic blood pressure; Test type: Superiority; p = 0.6610, Median test
Statistical Analysis 2: Comparison: Raphamin vs Placebo; Comparison for Visit 2/Systolic blood pressure; Test type: Superiority; p = 0.4884, Median test
Statistical Analysis 3: Comparison: Raphamin vs Placebo; Comparison for Visit 3/Systolic blood pressure; Test type: Superiority; p = 0.3494, Median test
Statistical Analysis 4: Comparison: Raphamin vs Placebo; Comparison for Visit 1/Diastolic blood pressure; Test type: Superiority; p = 0.9531, Median test
Statistical Analysis 5: Comparison: Raphamin vs Placebo; Comparison for Visit 2/Diastolic blood pressure; Test type: Superiority; p = 0.5506, Median test
Statistical Analysis 6: Comparison: Raphamin vs Placebo; Comparison for Visit 3/Diastolic blood pressure; Test type: Superiority; p = 0.8259, Median test

12. Secondary Outcome: Percentage of Patients With Clinically Relevant Abnormal Laboratory Findings.
Description: Outcome Measure is based on the Hematology, blood chemistry, and urinalysis parameters, which are beyond the reference values at the end of treatment.
Time Frame: Day 1 through day 7 of the treatment and observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Raphamin | Placebo
Number analyzed (Participants) | 206 | 214
Participants | 1 | 0
Statistical Analysis 1: Comparison: Raphamin vs Placebo; Test type: Superiority; p = 0.49, Fisher Exact

ADVERSE EVENTS:
Time Frame: Registration of AEs begins after the first dose of study drug and continues throughout the entire period of study therapy - 14 days.
Arm/Group | Raphamin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/214
Serious Adverse Events (participants affected / at risk) | 1/206 | 0/214
Other Adverse Events (participants affected / at risk) | 6/206 | 5/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raphamin (N=206) | Placebo (N=214)
Worsening flu (Infections and infestations) | 1 (1) | 0 (0) — Fever, nasal congestion, sore throat, weakness, dry cough. Hospitalization. Recovery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raphamin (N=206) | Placebo (N=214)
Adenoiditis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial superinfection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Increased percentage of monocytes (Investigations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0)
Flu (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04918771/Prot_SAP_000.pdf